CLINICAL TRIAL: NCT01934933
Title: A Multi-center, Open Label, Random Clinical Trial of Etanercept and Celecoxib Alone/Combined Treatment in Effectiveness and Safety of Active Ankylosing Spondylitis
Brief Title: Etanercept and Celecoxib Alone/Combined Treatment in Effectiveness and Safety of Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Department of Rheumatology, Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2013]2-93
Record Dates: First submitted 2013-08-17; First posted 2013-09-04 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Ankylosing Spondylitis
Keywords: inflammation; etanercept; celecoxib; ankylsoing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Inflammation | interventions — Celecoxib; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- celebrex (Active Comparator): celebrex capsule, 0.2 gram bid, 52 weeks
  Interventions: Drug: celebrex
- Enbrel (Active Comparator): etanercept injection, 25mg per injection, 50mg/week, 52 weeks
  Interventions: Drug: Enbrel
- Enbrel plus Celebrex (Active Comparator): 50mg/week Enbrel by hypodermic injection plus Celebrex 0.2 gram bid, 52 weeks
  Interventions: Drug: Enbrel plus Celebrex

INTERVENTIONS:
Drug: celebrex
  Other Names: celecoxib
  Arms: celebrex
Drug: Enbrel
  Other Names: etanercept
  Arms: Enbrel
Drug: Enbrel plus Celebrex
  Other Names: celecoxib plus etanercept
  Arms: Enbrel plus Celebrex

SUMMARY:
This is a multi-center, open label, randomized clinical trial of etanercept and celecoxib alone/combined treatment in effectiveness and safety on active ankylosing spondylitis (AS). Subjects will be randomly assigned in a 1:1:1 ratio to one of the three groups (celexocib 200mg bid, etanercept 50mg qw, etanercept plus Celecoxib group) for 54 weeks. Primary endpoints are the magnetic resonance imaging (MRI) Spondyloarthritis Research Consortium of Canada (SPARCC) score of sacroiliac(SI) joint and spine, as well as the Assessment of SpondyloArthritis International Society (ASAS)20 response rate at 52 weeks.

DETAILED DESCRIPTION:
A multi-center, open label, randomized clinical trial evaluating the effectiveness and safety of etanercept and celecoxib alone/combined treatment will be conducted on active ankylosing spondylitis (AS) patients. Disease activity is defined as fulfilling three aspects below: BASDAI ≥ 4 or ASDAS≥ 2.1；CRP>6 mg/L or ESR 28 mm/1st hour；more than 2 and less than 16 syndesmophyts between cervical spine and lumber spine detected by X-ray. All patients were randomly assigned in a 1:1:1 ratio to one of the three treatment groups：celecoxib 200mg bid，etanercept 50mg qw and combined therapy for 52 weeks. Primary endpoints are the magnetic resonance imaging (MRI) Spondyloarthritis Research Consortium of Canada (SPARCC) score of sacroiliac(SI) joint and spine, as well as the Assessment of SpondyloArthritis International Society (ASAS) 20 response rate at 52 weeks. Key secondary Endpoints include the modified Stoke Ankylosing Spondylitis Spine Score (mSASSS), Spondyloarthritis Research Consortium of Canada (SPRACC) SI joint structural score (SSS), BASDAI, ASDAS, ASAS40, ASAS70 and ASAS5/6 response rate at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years
* Meet 1984 NewYork modified criteria for AS
* BASDAI≥4 or ASDAS score ≥ 2.1
* CRP>6 mg/L or ESR>28 mm/h
* Syndesmophyte quantity ≥2 and <16 of spine
* Sexually active women of childbearing potential must agree and commit to use a medically accepted form of contraception
* No active or latent tuberculosis infection.

Exclusion Criteria:

* Pregnant or breastfeeding women
* current or previous history of psoriasis or inflammatory bowel disease.
* infection with clinical significance within 24 weeks before screening
* receipt any bio-agents treatment within 12 weeks before screening
* corticosteroids intra-articular injections in last 3 months before the trial
* Significant concurrent medical events including: Gastrointestinal ulcer, myocardial infarction within 12 months before the screening visit, unstable angina pectoris, congestive heart failure.
* Alcohol and drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
the SPARCC score of spine and SI joint | 52th weeks
  the MRI SPARCC score of spine and SI joint on 52th week
ASAS20 response rate | 52th week
  ASAS20 response rate on 52th week

SECONDARY OUTCOMES:
ASAS40 response rate | 52th week
  ASAS40 response rate on 52th week
ASAS70 response | 52th week
  ASAS70 response rate on 52th week
ASDAS | 52th week
  ASDAS major improvement ASDAS clinically important improvement on 52th week
mSASSS score of spine | 52th week
  the mSASSS score of spine on 52th week
Spondyloarthritis Research Consortium of Canada (SPRACC) SI joint structural score (SSS) | 52th week
  the MRI SPARCC SSS score of spine on 52th week

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Prof, Study Director — Department of Rheumatology ,Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tu L, Zhao M, Wang X, Kong Q, Chen Z, Wei Q, Li Q, Yu Q, Ye Z, Cao S, Lin Z, Liao Z, Lv Q, Qi J, Jin O, Pan Y, Gu J. Etanercept/celecoxib on improving MRI inflammation of active ankylosing spondylitis: A multicenter, open-label, randomized clinical trial. Front Immunol. 2022 Aug 26;13:967658. doi: 10.3389/fimmu.2022.967658. eCollection 2022. PMID 36091030